CLINICAL TRIAL: NCT00729209
Title: A Study of ARRY-371797 in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Array Biopharma, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Organization: Array BioPharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: ARRAY-797-103
Record Dates: First submitted 2008-08-04; First posted 2008-08-07 (Estimated); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — ARRY-371797

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- ARRY-371797 (Schedule 1) (Experimental)
  Interventions: Drug: ARRY-371797, p38 inhibitor; oral
- ARRY-371797 (Schedule 2) (Experimental)
  Interventions: Drug: ARRY-371797, p38 inhibitor; oral
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo; oral

INTERVENTIONS:
Drug: ARRY-371797, p38 inhibitor; oral — multiple dose, single schedule
  Arms: ARRY-371797 (Schedule 1); ARRY-371797 (Schedule 2)
Drug: Placebo; oral — matching placebo
  Arms: Placebo

SUMMARY:
This is a Phase 1 study, involving a 29-day treatment period, designed to evaluate the pharmacokinetics and the effectiveness of investigational study drug ARRY-371797 in treating rheumatoid arthritis in patients receiving stable doses of methotrexate, and to further evaluate the drug's safety. Approximately 30 patients from the US will be enrolled in this study.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosed with rheumatoid arthritis (RA) at least 3 months prior to study start based upon the American College of Rheumatology (ACR) 1987 Revised Criteria.
* On a stable weekly dose of both methotrexate (MTX) (10 - 25 mg/week inclusively; either oral or parenteral) and folate (≥ 5 mg weekly ) for ≥ 6 weeks prior to study start and is willing to continue on these regimens for the duration of the study.
* Meets the ACR 1991 Revised Criteria for Global Functional Status in RA, Class I, II, or III.
* Completed an appropriate washout period if treated with specified therapies.
* Patients may continue on specified stable background therapy for RA (doses should be stable for at least 6 weeks prior to the first dose of study drug, unless the patient stops due to documented disease improvement, with Sponsor approval).
* Additional criteria exist.

Key Exclusion Criteria:

* Diagnosis of any other inflammatory or non-inflammatory arthritis (e.g. spondyloarthritis; fibromyalgia, psoriatic arthritis, crystal-proven gout) that may interfere with disease activity assessments and/or clinically apparent osteoarthritis which would affect subsequent efficacy measures.
* Has received any of the following prior treatments:

  1. Within 4 weeks of first dose of study drug: anakinra (Kineret®), etanercept (Enbrel®);
  2. Within 8 weeks of first dose of study drug: infliximab (Remicade®), adalimumab (Humira®), leflunomide (Arava®);
  3. At any time: rituximab (Rituxan®), alemtuzumab (CamPath®), any experimental B cell targeting agents.
* Treatment with potent CYP3A inhibitors or inducers, disease-modifying antirheumatic drugs (DMARDs) and/or biologic response modifiers (BRMs) during the study.
* Additional criteria exist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2008-07; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Characterize the pharmacokinetics (PK) of the study drug and a metabolite in terms of plasma concentrations. | 29 days

SECONDARY OUTCOMES:
Characterize the safety profile of the study drug in terms of adverse events, clinical laboratory tests, vital signs and electrocardiograms. | 29 days
Assess the efficacy of study drug (versus placebo) in terms of cross-reactive protein (CRP), the Patient's Assessment of Arthritis Pain (100 mm visual analog scale [VAS]) and urinary N-Telopeptide Cross-Links (NTx). | 29 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (7):
- United States (7):
  - Clinic for Rheumatic Diseases, Tuscaloosa, Alabama
  - Sun Valley Arthritis Center, Ltd, Peoria, Arizona
  - Woodland International Research Group, Little Rock, Arkansas
  - NUCATS Institute, Northwestern University, Chicago, Illinois
  - Lynn Health Sciences Institute, Oklahoma City, Oklahoma
  - Metroplex Clinical Research Center, Dallas, Texas
  - Sentara Clinical Research Group, Norfolk, Virginia